CLINICAL TRIAL: NCT02231047
Title: 64N Nutraceutical for the Prevention of Childhood Diarrhea and Pneumonia in Low Resource Settings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: H2O Health and Agriculture LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H2O - BCO1
Record Dates: First submitted 2014-08-28; First posted 2014-09-03 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Diarrhea; Pneumonia
Keywords: Diarrhea; Pneumonia; Child, Preschool; Infant; Dietary Supplements; Colostrums; Developing Countries
MeSH Terms: conditions — Diarrhea; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 64N Nutraceutical (Experimental): Powdered 64N Nutraceutical 40 mg/kg/day mixed in 12 ounces of a culturally appropriate warm drink for 1 week (7 days).
  Interventions: Dietary Supplement: 64N Nutraceutical
- No 64N Nutraceutical (Sham Comparator): Culturally appropriate 12 ounce warm drink daily for 1 week (7 days).
  Interventions: Other: No 64N Nutraceutical

INTERVENTIONS:
Dietary Supplement: 64N Nutraceutical — 40 mg/kg/day of powdered 64N mixed in 12 ounces of a warm drink for 1 week (7 days)
  Other Names: Bovine colostrum
  Arms: 64N Nutraceutical
Other: No 64N Nutraceutical — 12 ounce warm drink daily for 1 week (7 days)
  Arms: No 64N Nutraceutical

SUMMARY:
The purpose of this study is to compare the occurrence of childhood diarrheal disease and pneumonia in subjects under the age of 5 years in low resource settings who have received prophylactic 64N nutraceutical (64N)as a neonate as compared with neonates who have not received prophylactic 64N.

DETAILED DESCRIPTION:
Diarrheal disease and pneumonia are two of the top four causes of mortality in children under the age of five . In 2010, 64 percent of deaths in this age group were due to infectious causes. A majority of these deaths occur in developing countries. Although vaccines have been proven to prevent pneumonia and diarrheal disease due to rotavirus, these vaccines may not be available to the most vulnerable children in developing countries. Barriers to vaccination in the poorest countries include lack of infrastructure, poor health systems, lack of finances, and lack of transportation. It has been estimated that an additional one billion US dollars will be needed to guarantee that the most vulnerable populations receive vaccinations.

Diarrheal disease is especially problematic since pathogens other than rotavirus cause diarrhea in children living in developing countries. Examples of pathogens causing diarrhea include Vibrio cholera, Salmonella enterica serovar Typhi, Escherichia coli [E. coli], Cryptosporidium, Entamoeba histolytica, and Shigella. Parasitic worms of the Schistosoma genus also cause diarrheal disease in poor countries. In developing countries, infants 0 to 11 months of age are at the highest risk of dying from diarrhea caused by typical E. coli and E. coli producing heat-stable toxin. Children 12 to 23 months of age are at the highest risk of dying from diarrhea caused by Cryptosporidium. It has been recommended that five pathogens (i.e., typical E. coli, E. coli producing heat-stable toxin, Cryptosporidium, Shigella, rotavirus) be targeted in order to decrease the burden of moderate-to-severe childhood diarrhea in developing countries.

In order to improve survival for children under the age of five in low resource settings, cost-effective, patient-directed, accessible, innovative, and alternative interventions that are culturally appropriate need to be explored. One such intervention that may confer passive immunity to protect young children in low resource settings against the multiple pathogenic causes of childhood diarrhea as well as childhood pneumonia is the utilization of 64N.

64N has been used by Ayurvedic physicians for medicinal purposes in humans in India and was also commonly used in Western medicine prior to the development of penicillin and other manufactured antibiotics. Both hyperimmune 64N and unadulterated 64N have been studied in children. Infants fed defatted hyperimmune 64N significantly decreased diarrhea due to rotavirus as compared with infants who received milk from the market. In children 3 to 15 months of age, 64N decreased rotavirus infection as compared with artificial infant formula.

Treatment studies have also shown a benefit of 64N for diarrhea. In children presenting with diarrhea due to E. coli, administration of 64N significantly decreased stool frequency as compared with placebo. 64N concentrates were found to be effective in the treatment of infants with hemorrhagic diarrhea and stopped the progression of the disease to hemolytic urea syndrome. 64N has also been studied in children (1 to 10 years of age) who had mild to moderate nonorganic failure to thrive. In this randomized controlled trial, the authors found that the Gomez index (a weight for age index) was significantly improved with 3 months of 64N supplementation as compared with no 64N supplementation.

There are few side effects of 64N. These are limited to lactose intolerance and sensitivity to milk proteins.

ELIGIBILITY:
Inclusion Criteria:

* Healthy neonates

Exclusion Criteria:

* Neonates with milk intolerance
* Neonates with lactose intolerance
* Premature neonates
* Neonates in poor health or who are being followed by a medical provider for illness

Ages: 6 Hours to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Mortality from childhood diarrhea and pneumonia | Assessed every 3 months for 4.5 years

SECONDARY OUTCOMES:
Medical visits for childhood diarrhea and pneumonia | Every 3 months for 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Donna M Rohrs, DHSc, PA, Principal Investigator — H2O Health and Agriculture LLC
Locations (1):
- Santa María de Jesús, Departamento de Sacatepéquez, Guatemala

REFERENCES:
- [Background] Ballard O, Morrow AL. Human milk composition: nutrients and bioactive factors. Pediatr Clin North Am. 2013 Feb;60(1):49-74. doi: 10.1016/j.pcl.2012.10.002. PMID 23178060
- [Background] Davidson GP, Whyte PB, Daniels E, Franklin K, Nunan H, McCloud PI, Moore AG, Moore DJ. Passive immunisation of children with bovine colostrum containing antibodies to human rotavirus. Lancet. 1989 Sep 23;2(8665):709-12. doi: 10.1016/s0140-6736(89)90771-x. PMID 2570959
- [Background] Ebina T, Sato A, Umezu K, Ishida N, Ohyama S, Oizumi A, Aikawa K, Katagiri S, Katsushima N, Imai A, et al. Prevention of rotavirus infection by oral administration of cow colostrum containing antihumanrotavirus antibody. Med Microbiol Immunol. 1985;174(4):177-85. doi: 10.1007/BF02123694. PMID 4069083
- [Background] Godhia, ML, Patel, N. Colostrum - its composition, benefits as a nutraceutical: A review. Current Research in Nutrition and Food Science, 1(1), 37-47, 2013.
- [Background] Huppertz HI, Rutkowski S, Busch DH, Eisebit R, Lissner R, Karch H. Bovine colostrum ameliorates diarrhea in infection with diarrheagenic Escherichia coli, shiga toxin-producing E. Coli, and E. coli expressing intimin and hemolysin. J Pediatr Gastroenterol Nutr. 1999 Oct;29(4):452-6. doi: 10.1097/00005176-199910000-00015. PMID 10512407
- [Background] Hurley WL, Theil PK. Perspectives on immunoglobulins in colostrum and milk. Nutrients. 2011 Apr;3(4):442-74. doi: 10.3390/nu3040442. Epub 2011 Apr 14. PMID 22254105
- [Background] Kotloff KL, Nataro JP, Blackwelder WC, Nasrin D, Farag TH, Panchalingam S, Wu Y, Sow SO, Sur D, Breiman RF, Faruque AS, Zaidi AK, Saha D, Alonso PL, Tamboura B, Sanogo D, Onwuchekwa U, Manna B, Ramamurthy T, Kanungo S, Ochieng JB, Omore R, Oundo JO, Hossain A, Das SK, Ahmed S, Qureshi S, Quadri F, Adegbola RA, Antonio M, Hossain MJ, Akinsola A, Mandomando I, Nhampossa T, Acacio S, Biswas K, O'Reilly CE, Mintz ED, Berkeley LY, Muhsen K, Sommerfelt H, Robins-Browne RM, Levine MM. Burden and aetiology of diarrhoeal disease in infants and young children in developing countries (the Global Enteric Multicenter Study, GEMS): a prospective, case-control study. Lancet. 2013 Jul 20;382(9888):209-22. doi: 10.1016/S0140-6736(13)60844-2. Epub 2013 May 14. PMID 23680352
- [Background] Liu L, Johnson HL, Cousens S, Perin J, Scott S, Lawn JE, Rudan I, Campbell H, Cibulskis R, Li M, Mathers C, Black RE; Child Health Epidemiology Reference Group of WHO and UNICEF. Global, regional, and national causes of child mortality: an updated systematic analysis for 2010 with time trends since 2000. Lancet. 2012 Jun 9;379(9832):2151-61. doi: 10.1016/S0140-6736(12)60560-1. Epub 2012 May 11. PMID 22579125
- [Background] Panahi Y, Falahi G, Falahpour M, Moharamzad Y, Khorasgani MR, Beiraghdar F, Naghizadeh MM. Bovine colostrum in the management of nonorganic failure to thrive: a randomized clinical trial. J Pediatr Gastroenterol Nutr. 2010 May;50(5):551-4. doi: 10.1097/MPG.0b013e3181b91307. PMID 20639714
- [Background] Solomons NW. Modulation of the immune system and the response against pathogens with bovine colostrum concentrates. Eur J Clin Nutr. 2002 Aug;56 Suppl 3:S24-8. doi: 10.1038/sj.ejcn.1601480. PMID 12142957
- [Background] Stelwagen K, Carpenter E, Haigh B, Hodgkinson A, Wheeler TT. Immune components of bovine colostrum and milk. J Anim Sci. 2009 Apr;87(13 Suppl):3-9. doi: 10.2527/jas.2008-1377. Epub 2008 Oct 24. PMID 18952725
- [Background] Struff WG, Sprotte G. Bovine colostrum as a biologic in clinical medicine: a review--Part II: clinical studies. Int J Clin Pharmacol Ther. 2008 May;46(5):211-25. doi: 10.5414/cpp46211. PMID 18538107
- [Background] World Health Organization. Causes of child mortality, by region, 2000-2011. In Global health observatory (GHO), (2014) Retrieved from http://www.who.int/gho/child_health/mortality/mortality_causes_region_text/en/
- [Background] World Health Organization. Childhood vaccines at all-time high, but access not equitable, (2009). Retrieved from http://www.who.int/mediacentre/news/releases/2009/state_immunizaton_200910